CLINICAL TRIAL: NCT06428240
Title: Reality of Acute Mesenteric Ischemia in Catalonia, is There a Chance to Improvement?
Brief Title: Acute Mesenteric Ischemia, Reality in Catalonia
Acronym: AMI_CAT
Status: Not yet recruiting | Type: Observational
Sponsor: Hospital del Mar (Other)
Collaborators: Hospital Clinic of Barcelona (Other); Germans Trias i Pujol Hospital (Other); Parc Taulí Hospital Universitari (Other); Hospital de la Santa creu i Sant Pau - Barcelona (Other); Hospital Vall d'Hebron (Other); Hospital Universitari Joan XXIII de Tarragona. (Other); Hospital de Manresa (Unknown); Hospital de Mataró (Other); Hospital Universitari Sant Joan de Reus (Other); Hospital de Sant Joan Despí Moisès Broggi (Other); Hospital d'Igualada (Other); Consorci Hospitalari de Vic (Other); Hospital Arnau de Vilanova (Other); Hospital de Mollet (Unknown); Hospital de Terrassa (Other); Hospital Universitari de Bellvitge (Other)
Responsible Party: Principal Investigator, Ana María González Castillo, Doctor, Hospital del Mar
Other Study IDs: AMICat Reality
Record Dates: First submitted 2024-05-20; First posted 2024-05-24 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Acute Mesenteric Ischemia
Keywords: Mesenteric ischemia; Acute Mesenteric ischemia; Abdominal pain; Elderly; Complications; Mortality
MeSH Terms: conditions — Mesenteric Ischemia; Abdominal Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Acute mesenteric ischaemia (AMI) is a notorious disease with a high mortality, the diagnostic and management is truly multidisciplinary, but not very extended. The aim of this study is to analyse the results of the patients admited with an AMI in Catalonia.

DETAILED DESCRIPTION:
Acute mesenteric ischaemia (AMI) is a notorious disease with a high mortality from 50 to 80%. Even though AMI is a relatively rare condition (1:1,000) the incidence rises exponentially with increasing age, in patients older than 75 years, the incidence of AMI has been reported higher than that of acute appendicitis. AMI patients benefit from early assessment in a surgical unit with capabilities to definitive management. The diagnosis and management of AMI are truly multidisciplinary, requiring high index of suspicion and awareness from emergency department physicians, preferably computed tomography angiography with precise interpretation, but usually this is not the truth reality and the diagnostic is delayed as well as the treatment, and the management is not multidisciplinary.

The aim of this study is to analyse the management and results of the patients admitted with an AMI in Catalonia from November 2024 to April 2026.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic of Acute Mesenteric Ischemia

Exclusion Criteria:

* Chronic Mesenteric Ischemia
* Ischemic Colitis
* Bowel obstruction strangulation
* Inflammatory bowel necrosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: The study populations is all pacients with the diagnostic of Acute Mesenteric Ischemia that are admitted in the Hospital in Catalonia.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2024-11-01 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Mortality | 2024-2026
  To describe the mortality in patients with a diagnostic of AMI

SECONDARY OUTCOMES:
Complications | 2024-2026
  To describe the complications in patients with a diagnostic of AMI
Management | 2024-2026
  To describe the management in patients with a diagnostic of AMI